CLINICAL TRIAL: NCT01465685
Title: Emotional Effects of Methylphenidate and MDMA in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 228/11
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: MDMA; pharmacokinetics; pharmacodynamics; emotions; Mechanism of action of MDMA; Interaction study; Effect of MDMA and methylphenidate on emotions
MeSH Terms: interventions — N-Methyl-3,4-methylenedioxyamphetamine; Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDMA, methylphenidate, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject.
  Interventions: Drug: 3,4-Methylenedioxymethamphetamine; Drug: Methylphenidate; Drug: Placebo

INTERVENTIONS:
Drug: 3,4-Methylenedioxymethamphetamine — 125 mg per os, single dose
  Other Names: MDMA; ecstasy
Drug: Methylphenidate — 1 hour before MDMA/placebo 60 mg methylphenidate per os, single dose
  Other Names: Ritalin; Concerta
Drug: Placebo — capsules identical to MDMA or methylphenidate

SUMMARY:
This study compares the interactive emotional/subjective effects of single doses of 3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") and methylphenidate, a dopamine (DA) and norepinephrine (NE) transporter blocker, in healthy subjects. The primary goal is to determine the role of transporter mediated DA and NE release in the subjective response to MDMA in humans. The investigators hypothesize that methylphenidate will attenuate the subjective response to MDMA.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), dopamine (DA), and norepinephrine (NE). 5-HT release mainly contributes to the subjective effects of MDMA whereas NE release is involved in the cardiovascular and psychostimulant effects of MDMA. DA is also likely to be involved in the rewarding and reinforcing effects of drugs of abuse. However, the functional role of DA in the subjective effects of MDMA in humans is largely unclear. To determine the role of the DA transporter (DAT) in the response to MDMA in humans the investigators test the effects of the DA and NE transporter blocker methylphenidate on the subjective effects of MDMA. The investigators use a randomized double-blind placebo-controlled cross-over design with four experimental sessions. methylphenidate or placebo will be administered before MDMA or placebo to 16 healthy volunteers. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics. The primary hypothesis is that methylphenidate will significantly reduce the subjective effects of MDMA.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to refrain from taking illicit psychoactive substances during the study.
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing liquids (such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session. Subjects must agree not to smoke tobacco for 1 h before and 4 hours after MDMA administration.
* Participants must be willing not to drive a traffic vehicle in the evening of the study day.
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session.
* Body mass index: 18-25 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder.
* Current or previous psychotic or affective disorder
* Psychotic or affective disorder in first-degree relatives
* Prior illicit drug use (except THC-containing (tetrahydrocannabinol) products) more than 5 times or any time within the previous 2 months.
* Pregnant or nursing women.
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Subjective effect during 24 hours | 24 hours
  subjective effects are repetitively assessed by standardized questionnaires.

SECONDARY OUTCOMES:
Blood pressure (mmHg)during 10 hours | 10 hours
Neuroendocrine plasma levels during 10 hours | 10 hours
  neuroendocrine parameters assessed: prolactin, cortisol, epinephrine, norepinephrine, oxytocin, pro-vasopressin, vasopressin, estrogen,and progesterone
MDMA plasma levels during 24 hours | 24 hours
Heart rate (beats/min)) during 10 hours | 10
Emotional and cognitive empathy | 5 hours
  emotional empathy is going to be assessed by the Multifaceted Empathy Test (MET).
  cognitive empathy is going to be assessed by the Facial Emotion Recognition Task and the MET.
Prosocial behavior | 5 hours
  Effects on prosociality will be assessed by the Social Value Orientation slide-measurement test.
Genetic polymorphisms | assessed after study completion
  Effects of genetic polymorphisms on the response to MDMA

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Hysek CM, Simmler LD, Schillinger N, Meyer N, Schmid Y, Donzelli M, Grouzmann E, Liechti ME. Pharmacokinetic and pharmacodynamic effects of methylphenidate and MDMA administered alone or in combination. Int J Neuropsychopharmacol. 2014 Mar;17(3):371-81. doi: 10.1017/S1461145713001132. Epub 2013 Oct 8. PMID 24103254